CLINICAL TRIAL: NCT04357509
Title: An Open-lable,Single-arm,Single-dose Escalation and Multiple-dose Expansion Clinical Study of Cell Therapy to Observe and Evaluate the Tolerance,Pharmacokinetic Characteristics,Safety and Efficacy of ScTIL210 in the Treatment of Melanoma
Brief Title: The Tolerance,Pharmacokinetic Characteristics,Safety and Efficacy of ScTIL210 in the Treatment of Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScTIL210-002-2019
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ScTIL210 (Experimental): This trial is designed single arm. All the subjects enrolled will receive the experimental intervention, ScTIL210(Super circulating tumor infiltrating lymphocytes).
  Interventions: Biological: Super circulating tumor infiltrating lymphocytes(ScTIL)

INTERVENTIONS:
Biological: Super circulating tumor infiltrating lymphocytes(ScTIL) — Peripheral blood mononuclear cells (PBMCs) are used for cell preparation. PD-1(programmed death 1) positive T cells are isolated from peripheral blood by blood cell apheresis method and transduced with lentivirus loaded with "enhanced receptor" and "superamplification factor". The obtained ScTIL is used for one-time intravenous infusion.

SUMMARY:
This is an open-lable, single-arm, single-dose escalation and multiple-dose expansion clinical study of cell therapy to observe and evaluate the tolerance, pharmacokinetic characteristics, safety and efficacy of ScTIL210（Super circulating tumor infiltrating lymphocytes）in the treatment of Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old (inclusive), regardless of gender.
2. Expected survival duration is greater than three months.
3. Patients with acral and mucosal melanoma confirmed by histology or cytology.
4. Disease progression after previous first-line system treatment or intolerance during the treatment. Intolerance includes the following:

   1. Incompetence of major organ function restoration of the subject as judged by the investigator.
   2. The subjects experienced Grade 3 non-hematological toxicity or Grade 4 hematological toxicity during treatment (Grade 3 thrombocytopenia).
   3. The subjects refuse the optional first-line treatment.
5. Subjects voluntarily accept peripheral blood apheresis to obtain cells for cell preparation. The proportion of peripheral blood PD1(programmed death 1)positive T cells in total T cells is ≥18%. The proportion of peripheral blood PD1 positive T cells in total T cells ratio is ≥12% for the subjects underwent PD1 monoclonal antibody treatment before screening.
6. At least one measurable focal lesion (for efficacy assessment) has been detected by CT or MRI as defined by RECIST v1.1. The measurable tumor lesion is defined as the longest diameter ≥ 10mm and the short diameter of metastatic lymph nodes ≥ 15mm under the condition that the scanning thickness does not exceed 5.0 mm;
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. No serious hematology, liver, and kidney dysfunction, and meet the following laboratory test criteria:

   1. Hematology: neutrophils is equal to or higher than 1.5×10^9/L, platelets is equal to or higher than 75×10^9/L, hemoglobin is equal to or higher than 90g/L; total lymphocytes is equal to or higher than 50% of the normal lower line;
   2. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are both eqal to or lower than 3 times the upper limit of normal (ULN) (if intrahepatic bile duct cancer exists, equal to lower than 5 times of ULN); total bilirubin (TBIL) is equal to or lower than 2 times of ULN;
   3. Kidney function: creatinine (Cr) is equal to or lower than 1.5 times of ULN;
   4. Coagulation function: prothrombin time (PT) is equal to or shorter than 1.5 times of ULN or activated partial prothrombin time (APTT) is equal to or shorter than1.5 times of ULN;
   5. Urine protein concentration is equal to or lower than ≤ 1 +, no edema.
   6. Albumin is equal to or higher than 3.0g/dl.
9. At the beginning of screening, the elution period upon completion of anticancer chemotherapies and glucocorticoids (includes hydrocortisone, prednisone, prednisolone, methylprednisolone) should be no shorter than 4 weeks; Palliative radiotherapy is allowed, as long as the selected region(s) of the therapy is/are spatially distinct from that correspondent to designated focus of lesion for efficacy assessment.
10. Male or fertile female subjects are required to take effective contraceptive measures during the treatment as well as within 90 days upon completion of last therapeutic cell reinfusion;
11. Full capability and commitment to abide by clinical research protocols and follow-up procedures.
12. Subjects understand and are willing to abide by the study protocol and to participate in the study by providing signed informed consent form.

Exclusion Criteria:

1. Subjects with Uveal/Ocular melanoma.
2. Subjects with symptomatic and/or untreated brain metastases (of any size and number).

   a) Subjects with treated brain metastases can be considered for enrollment under the condition that the disease must have remained stable for greater than 14 days before starting screening.
3. Subjects with another primary malignancy within the past 3 years including breast cancer, cervical cancer, bladder cancer in situ, and local prostate cancer);
4. Presence of any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; with exclusion of Asthma subjects who need bronchodilators for medical intervention); however, the following patients are allowed:

   1. Vitiligo, psoriasis, hair loss without systemic treatment;
   2. Well-controlled type 1 diabetes;
   3. Hypothyroidism with replacement thyroid function.
5. Subjects receiving chronic systemic steroid treatment for any reason; with exception of the low-dose glucocorticoid replacement therapy due to adrenal insufficiency.
6. Recipients of any organ transplant, including allogeneic stem cell transplants, with exception of transplants requiring no immunosuppression (e.g, corneal transplants, hair transplants).
7. Subjects with any forms of primary immunodeficiency (e.g, severe combined immunodeficiency disease [SCID] and acquired immunodeficiency syndrome [AIDS])
8. Presence of major acute or chronic infections, including:

   1. A known history of positive human immunodeficiency virus (HIV) or a known history of acquired immunodeficiency syndrome (not required for screening). If the investigator strongly suspects a HIV infection in a subject with no known medical history during the screening period, the subject should be tested for HIV in accordance to the local standard guidelines).
   2. Active TB infection (evidences are: clinical symptoms, physical examination and/or medical imaging, and laboratory findings).
   3. An active bacterial or fungal infection that requires systemic treatment.
   4. Viral hepatitis, including hepatitis B and C, etc.
   5. Subjects with syphilis virus positive
9. Acute exacerbation of chronic obstructive pulmonary disease , or other respiratory diseases that requires hospitalization within 30 days prior to enrollment，or that hinders study treatment.
10. Clinically significant cardiovascular or cerebrovascular diseases, such as: cerebrovascular accident or stroke occured within6 months prior to enrollment), myocardial infarction (occured within6 months prior to enrollment), unstable angina, congestive heart failure (equal to or greater than Grade II of New York Heart Association) or severe arrhythmia.
11. Subjects who are incapable tolerate or are allergic to contrast agents of CT scanning or magnetic resonance imaging (MRI).
12. Subjects who participated in other clinical trials within 4 weeks prior to enrollment.
13. Pregnant or lactating women.
14. A history of alcoholic or drug abuse within 2 years (acknowledged via inquiries and previous medical history) prior to enrollment.
15. Other severe acute or chronic diseases, or incompetency/have only restricted competency for civil conduct.
16. Subjects or family members is/are incapable to understand the conditions and goals of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 24 weeks after the last cell transfusion
  Including cases of CR and PR

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | 24 weeks after the last cell transfusion
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases
Duration of Response(DOR) | 24 weeks after the last cell transfusion
  Time from complete remission (CR) or partial remission (PR) to disease progression (PD), death or last tumor evaluation
Progression-Free Survival(PFS) | 24 weeks after the last cell transfusion
  From the beginning of cell therapy to the time of the first disease progression or death due to any cause
Overall survival(OS) | 24 weeks after the last cell transfusion
  Time from cell reinfusion to death due to any cause
Adverse events(AEs) | 24 weeks after the last cell transfusion
  According to National Cancer Institute Common Terminology Criteria for Adverse Events V5.0(CTCAE V5.0)
Detection of Lentivirus Copy Number | 24 weeks after the last cell transfusion
  Dynamic changes of carrier gene copy number in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China